CLINICAL TRIAL: NCT03087669
Title: Evaluation of Central and Cerebral Circulation in Early Stages After Implantation of Left Ventricular Assist Device (LVAD)
Brief Title: Central and Cerebral Circulation in Early Stages After LVAD Implantation
Acronym: ECOH3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bjorn Reinsfelt, Head of Department of Cardiac Anesthesia. Consultant. PhD, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECOH 3
Record Dates: First submitted 2017-02-28; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure, Left-Sided; Heart Failure, Right-Sided
Keywords: Left Ventricular Assist Device; Hemodynamic monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: 1. LVAD will have a setting of 4800 rounds per minute (RPM). Hemodynamic, echocardiographic and cerebral blood flow measurements will be performed: CO, PCWP, CVP, PAP, MAP, Peripheral and central hemoglobine oxygen saturation (SaO2 and SvO2), Heart Rate (HR), RV outflow tract Velocity Time Integral (RVOT VTI), RV and LV diameter, VTI of LVAD outflow. CBFV of right and left medial cerebral artery (RMCA and LMCA)
  2. The above mentioned measurements will be repeated with LVAD settings of 5200 RPM, 5600 RPM, and 6000 RPM.
  3. With the LVAD fixed to an optimized setting detected by the previous interventions, the blood pressure will be adjusted to MAP 60 mmHg. The above mentioned measurements will be repeated.
  4. Using Noradrenaline the MAP will be adjusted to 70mmHg, 80 mmHg and 90 mmHg. At steady state for each level of MAP with a fixed LVAD flow, all the above mentioned measurements will be repeatedly performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation of hemodynamic parameters (Experimental): LVAD flow velocity setting-Rounds Per Minute(RPM) intervention: Change of LVAD RPM while observing Central hemodynamic, echocardiographic and CBFV effects.
  MAP intervention: Stepwise Change of MAP from 60-70-80 to 90 mmHg with a fixed set of LVAD RPM. After a 5 minute steady state for each level of MAP, the observations of central hemodynamics, echocardiographic measures and CBFV measurements will be repeated.
  Interventions: Device: LVAD flow velocity setting-Rounds per Minute(RPM) on HeartMate III®; Drug: MAP intervention using Noradrenalin

INTERVENTIONS:
Device: LVAD flow velocity setting-Rounds per Minute(RPM) on HeartMate III® — Increase in LVAD RPM setting induces an actual increase in LVAD outflow to the patient.This gives the patient an increased systemic Cardiac Output(CO)
  Other Names: RPM setting
Drug: MAP intervention using Noradrenalin — At a fixed RPM rate for the LVAD the Mean Arterial Pressure (MAP) is increased to preset levels of 60-70-80-90 mmHG using Noradrenalin
  Other Names: MAP setting

SUMMARY:
This trial will evaluate patients with a mechanical Left Ventricular Assist Device (LVAD) in early stages after surgical implantation. Within the first 2 days of postoperative ICU care, 20 patients will firstly be exposed to 4 different LVAD pump flow settings with a stable blood pressure. A second intervention will be mean arterial blood pressure (MAP) adjustments to 4 preset levels (60-70-80 and 90 mmHg) with a constant preset LVAD flow. The two manipulations; 1) Constant MAP with variation of LVAD flow and 2) Constant LVAD flow with variation of MAP, will be monitored by Central hemodynamic parameters, echocardiographic parameters and cerebral blood flow velocity (CBFV) parameters. The purpose of the trial is to find the optimal combination of LVAD pump flow, mean arterial pressure and right heart ventricle function for each patient. And at the same time describe the effect of flow and pressure variations on CBFV.

DETAILED DESCRIPTION:
Patients with severe left ventricular heart failure and estimated short expected survival time despite optimal medical therapy can be treated with a left ventricular mechanical heart pump - described as a Left Ventricular Assist Device (LVAD). The LVAD can be used as a bridge for patient survival prior to heart transplantation, or as a destination therapy for terminal heart failure. The LVAD delivers a non-pulsatile blood flow into the patients aorta, supporting and/or taking over the left ventricular function. However the right heart ventricle (RV) is not supported by the LVAD. RV failure is a major threat to the patient, in particular during the early postoperative period. Postoperative RV failure after LVAD implantation is medically treated, but in severe cases a mechanical temporary right ventricular assist (RVAD) may be needed. Patients in need of postoperative RVAD after an LVAD implant have a significantly increased mortality. Thus it is of vital importance to balance the LVAD pump flow against the native RV function in order to avoid the need for an RVAD. If the LVAD flow rate is set too low the RV will be exposed to a high afterload and risk failure. If, on the other hand, the LVAD flow is set too high it can potentially completely empty the left ventricle with secondary geometrical distortion of the heart chambers and an increased venous return to the RV. This too increases the risk for RV failure. To find the optimal LVAD flow rate it is custom to do an extensive evaluation of central hemodynamic parameters (Cardiac Output(CO), Pulmonary Capillary Wedge Pressure (PCWP), Pulmonary Arterial Pressure (PAP), Central Venous Pressure (CVP)) and cardiac echocardiographic evaluation of RV function at different LVAD pump flow rates and MAP. The instant balance between RV filling pressure-CVP, and LV filling pressure-PCWP, is on the other hand easy to obtain. However it is not known if these measurements can be used to obtain an optimal LVAD flow rate. Furthermore all mechanically driven circulatory support devices, including LVAD, will expose the peripheral arterial circulation to a non-pulsatile blood flow.There are few previous reports on how an LVAD affects the cerebral blood flow autoregulation and microembolic load at different settings and MAP. This investigation aims to describe these cerebral effect af an LVAD using a continous Transcranial Doppler (TCD) detection of cerebral arteries.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving LVAD of the type HeartMate3® at Sahlgrenska University hospital

Exclusion Criteria:

* Perioperative need for an RVAD first 3 days postoperatively after an LVAD implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes PCWP/CVP ratio | Change from baseline at different settings of LVAD RPM within 10 minutes for each level
  The change in PCWP (mmHg)/CVP (mmHg) ratio at different levels of LVAD flow as a marker for the optimal balance between LVAD flow and RV function

SECONDARY OUTCOMES:
CO | Change from baseline at different settings of LVAD RPM within 10 minutes for each level
  Cardiac Output in litres/minute
LVAD Velocity Time Integral | Change from baseline at different settings of LVAD RPM within 10 minutes for each level
  LVAD Velocity Time Integral in centimeters(cm)
Right Ventricle Outflow Tract (RVOT) Velocity Time Integral (VTI) | Change from baseline at different settings of LVAD RPM within 10 minutes for each level
  RVOT Velocity Time Integral in centimeters(cm)
CBFV | Change from baseline at different settings of LVAD RPM within 10 minutes for each level
  CBFV in cm/second

OTHER OUTCOMES:
Changes PCWP/CVP ratio at different MAP | Change from baseline at different settings of MAP with a fixed LVAD RPM setting within 10 minutes for each level
  The change in PCWP (mmHg)/CVP (mmHg) ratio at different levels of MAP as a marker for the optimal balance between LVAD flow and RV function
LVAD VTI at different MAP | Change from baseline at different settings of MAP with a fixed LVAD RPM setting within 10 minutes for each level
  LVAD Velocity Time Integral in centimeters(cm)
CO at different MAP | Change from baseline at different settings of MAP with a fixed LVAD RPM setting within 10 minutes for each level
  Cardiac Output in litres/minute
RVOT VTI at different MAP | Change from baseline at different settings of MAP with a fixed LVAD RPM setting within 10 minutes for each level
  RVOT Velocity Time Integral in centimeters(cm)
CBFV at different MAP | Change from baseline at different settings of MAP with a fixed LVAD RPM setting within 10 minutes for each level
  CBFV in cm/second

CONTACTS AND LOCATIONS:
Overall Officials: Sven Erik Ricksten, MD.PhD, Study Director — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital. Department of Cardiothoracic Anaesthesia & Intensive Care, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uriel N, Adatya S, Maly J, Kruse E, Rodgers D, Heatley G, Herman A, Sood P, Berliner D, Bauersachs J, Haverich A, Zelizko M, Schmitto JD, Netuka I. Clinical hemodynamic evaluation of patients implanted with a fully magnetically levitated left ventricular assist device (HeartMate 3). J Heart Lung Transplant. 2017 Jan;36(1):28-35. doi: 10.1016/j.healun.2016.07.008. Epub 2016 Jul 17. PMID 27773456
- [Result] Uriel N, Sayer G, Addetia K, Fedson S, Kim GH, Rodgers D, Kruse E, Collins K, Adatya S, Sarswat N, Jorde UP, Juricek C, Ota T, Jeevanandam V, Burkhoff D, Lang RM. Hemodynamic Ramp Tests in Patients With Left Ventricular Assist Devices. JACC Heart Fail. 2016 Mar;4(3):208-17. doi: 10.1016/j.jchf.2015.10.001. Epub 2015 Dec 30. PMID 26746378
- [Result] Ono M, Joshi B, Brady K, Easley RB, Kibler K, Conte J, Shah A, Russell SD, Hogue CW. Cerebral blood flow autoregulation is preserved after continuous-flow left ventricular assist device implantation. J Cardiothorac Vasc Anesth. 2012 Dec;26(6):1022-8. doi: 10.1053/j.jvca.2012.07.014. PMID 23122299